CLINICAL TRIAL: NCT04007679
Title: The Effects of Pain Neuroscience Education in Undergraduate Physiotherapy
Brief Title: Pain Neuroscience Education in Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principal Investigator, Kutahya Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KutahyaMSUnpq
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain; Educational Problems
Keywords: pain neuroscience education; chronic pain; physiotherapy students
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pain education group (Experimental): Pain education was conducted in physical conditions similar to the university classrooms where the study was performed for all participants.
  Interventions: Other: Pain neuroscience education

INTERVENTIONS:
Other: Pain neuroscience education — Pain neuroscience education (PNE) was conducted in physical conditions similar to the university classrooms where the study was performed. The sessions were conducted as 70-minute didactic group lessons with the same content held in separate sessions for students in each class. PowerPoint (Microsoft Corp., Redmond, WA, USA) presentations prepared by the instructor were used in all sessions. Metaphors, anecdotes, graphics, and pictures were used in an attempt to convey the information and messages about pain physiology and theory more permanently and effectively. In the PNE sessions, it was explained that the nervous system can be overprotective and that in addition to the sensitivity of the central nervous system, nociceptive transmission can be affected by an individual's thoughts, beliefs, and surroundings. At the end of the session, the students were given time to ask questions, but group discussion was limited to 15 minutes due to time restrictions.

SUMMARY:
This study was designed to evaluate the effect of a 70-minute Pain neuroscience education (PNE) session on physiotherapy students' knowledge of pain and their beliefs and attitudes about the treatment of patients with chronic pain.

DETAILED DESCRIPTION:
To investigate the effect of a 70 minute pain neuroscience education session on physiotherapy students' knowledge of pain and their beliefs and attitudes about the treatment of patients with chronic pain. This study was a single-center, cross-sectional study on the pain knowledge of students in a four-year physiotherapy program and their beliefs and attitudes about patients with back pain.Students were eligible to participate if they were enrolled at physiotherapy undergraduate program at Kütahya Health Sciences University Faculty of Health Sciences. Individuals were excluded if they had previously received in depth-teaching on pain neuroscience. The study was completed with 156 students from different classes (first, second, and third year of the program) who agreed to participate in the study. All participants were informed about the study and signed informed consent forms. Pain neurophysiology questionnaire and Pain Attitudes and Beliefs Scale for Physiotherapists were used to assess pain knowladge and attitudes and beliefs. After recording their demographic information, the participants completed the Neuroscience of Pain Questionnaire (NPQ) and Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT) at three time points: pre-PNE, immediately post-PNE, and 6 months after PNE.

ELIGIBILITY:
Inclusion Criteria:

* participants who study in physiotherapy.
* willing to participate

Exclusion Criteria:

* Individuals in years 4 were excluded.
* participants who received an in-depth session about pain previously.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Neurophysiology of Pain Questionnaire (NPQ) | Baseline and six months
  The NPQ was designed to assess pain knowledge and consists of 19 questions with choices of "true", "false", or "I don't know." The questionnaire was developed in 2003 by Moseley , the validity study was conducted by Catley et al. , and it was determined as effective in the evaluation of pain knowledge. The total score is 0-19, with higher score indicating more correct answers. It was reported that the NPQ can be used both with healthcare professionals and with patients after some modifications to make it more comprehensible for patients.

SECONDARY OUTCOMES:
Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT) | Baseline and six months
  This tool was developed to distinguish between biomedical and biopsychosocial orientations toward the treatment of low back pain in physiotherapists. In the biomedical treatment orientation, the predominant belief is that the source of pain and disability is a specific pathology and tissue damage, and therefore the main goal is to treat the signs and symptoms of the pathology [19]. In the biopsychosocial treatment orientation, pain and disability can occur in the absence of tissue injury and are affected by psychological and social factors. The scale uses a 6-point Likert-type scale (1=definitely disagree, 6=definitely agree). Treatment orientation is measured on the biomedical (factor 1) and biopsychosocial (factor 2) subscales. Subscale scores are calculated by simply adding the scores corresponding to the selected response for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Cihan AKSOY, Phd, Study Director — Kutahya Health Sciences University
Locations (1):
- KutahyaMSU, Kütahya, Kutahya Health Sciences University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No